CLINICAL TRIAL: NCT00198003
Title: Addressing Patients Expectations of Total Hip Arthroplasty: Developing and Testing an Educational Intervention in a Randomized Trial
Brief Title: Addressing Patients' Expectations of Total Hip Arthroplasty in a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 99104
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Hip Osteoarthritis; Arthroplasty, Replacement, Hip
Keywords: hip arthritis; total hip arthroplasty; expectations; education
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Educational program to address patients' expectations

SUMMARY:
The goals of this study are to develop and test an educational intervention to address patients' expectations of long-term outcomes of total hip arthroplasty.

DETAILED DESCRIPTION:
The first goal of this study is to develop an educational intervention to address patients' expectations of long-term outcomes of total hip arthroplasty. The intervention will be structured according to the expectations listed in the Hospital for Special Surgery Total Hip Replacement Expectations Survey. The second goal is to test the intervention in a randomized trial. An additional goal is to compare patients' self-reported hip symptoms with radiographic findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for this study if they are 55 years of age or older and are scheduled for primary total hip arthroplasty at the Hospital for Special Surgery.

Exclusion Criteria:

* Patients will be excluded from this study for the following reasons: if they are not fluent in English; if they are not going to attend the preoperative hip replacement class; if they are unable to complete the surveys; if they refuse to participate.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2001-11; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the within-patient change between pre and post program scores measured by the Hospital for Special Surgery Total Hip Replacement Expectations Survey.

SECONDARY OUTCOMES:
The secondary outcome is to compare patient-reported symptoms with radiographic ratings of disease activity.
The secondary outcome is to assess if patients' expectations after the class coincide with orthopedic surgeons expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Mancuso CA, Sculco TP, Salvati EA. Patients with poor preoperative functional status have high expectations of total hip arthroplasty. J Arthroplasty. 2003 Oct;18(7):872-8. doi: 10.1016/s0883-5403(03)00276-6. PMID 14566742
- [Background] Mancuso CA, Ranawat CS, Esdaile JM, Johanson NA, Charlson ME. Indications for total hip and total knee arthroplasties. Results of orthopaedic surveys. J Arthroplasty. 1996 Jan;11(1):34-46. doi: 10.1016/s0883-5403(96)80159-8. PMID 8676117
- [Background] Blake VA, Allegrante JP, Robbins L, Mancuso CA, Peterson MG, Esdaile JM, Paget SA, Charlson ME. Racial differences in social network experience and perceptions of benefit of arthritis treatments among New York City Medicare beneficiaries with self-reported hip and knee pain. Arthritis Rheum. 2002 Aug;47(4):366-71. doi: 10.1002/art.10538. PMID 12209481
- [Background] Peterson MG, Hollenberg JP, Szatrowski TP, Johanson NA, Mancuso CA, Charlson ME. Geographic variations in the rates of elective total hip and knee arthroplasties among Medicare beneficiaries in the United States. J Bone Joint Surg Am. 1992 Dec;74(10):1530-9. PMID 1469013
- [Background] Mancuso CA, Salvati EA, Johanson NA, Peterson MG, Charlson ME. Patients' expectations and satisfaction with total hip arthroplasty. J Arthroplasty. 1997 Jun;12(4):387-96. doi: 10.1016/s0883-5403(97)90194-7. PMID 9195314
- [Result] Mancuso CA, Graziano S, Briskie LM, Peterson MG, Pellicci PM, Salvati EA, Sculco TP. Randomized trials to modify patients' preoperative expectations of hip and knee arthroplasties. Clin Orthop Relat Res. 2008 Feb;466(2):424-31. doi: 10.1007/s11999-007-0052-z. Epub 2008 Jan 10. PMID 18196427
- [Result] Mancuso CA, Pavlov H, Hays PL, Sculco TP. Symptoms associated with compartmental radiographic disease in hip arthroplasty patients. J Arthroplasty. 2011 Apr;26(3):439-44. doi: 10.1016/j.arth.2010.01.005. Epub 2010 Mar 23. PMID 20334992